CLINICAL TRIAL: NCT06145165
Title: A Analgesic Study of Adductor Canal &IPACK Block with Liposomal Bupivacaine in Knee Arthroplasty ：A Randomized，Double-controlled，Parallel-controlled，Single-center Study
Brief Title: A Analgesic Study of Adductor Canal &IPACK Block with Liposomal Bupivacaine in Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20230829-05
Record Dates: First submitted 2023-10-27; First posted 2023-11-24 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-11

CONDITIONS: Liposomal Bupivacaine; Postoperative Recovery; Unilateral Knee Arthroplasty
MeSH Terms: interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RP group:Nerve block with ropivacaine and intravenous analgesia group (Placebo Comparator): The ropivacaine group will use ultrasound high-frequency line array probe for ACB and convex array probe for iPACK block before induction of general anesthesia
  Interventions: Other: Nerve block with ropivacaine and intravenous analgesia
- LP group ：Nerve block with liposomal bupivacaine and intravenous analgesia group (Experimental): The liposomal bupivacaine group will use ultrasound high-frequency line array probe for ACB and convex array probe for iPACK block before induction of general anesthesia
  Interventions: Combination Product: Nerve block with liposomal bupivacaine and intravenous analgesia
- control group：Intravenous analgesia group (Placebo Comparator): General anesthesia was induced directly
  Interventions: Other: Intravenous analgesia

INTERVENTIONS:
Other: Nerve block with ropivacaine and intravenous analgesia — When the MOAA/S score is 5 after the surgery,the PCIA pump equipped with sufentanil injection will be connected,if the patient's resting NRS ≥ 4 points , they should be given sufentanil 5 ug intravenously at intervals of more than 8 minutes until NRS ≤ 3.
  Arms: RP group:Nerve block with ropivacaine and intravenous analgesia group
Combination Product: Nerve block with liposomal bupivacaine and intravenous analgesia — When the MOAA/S score is 5 after the surgery,the PCIA pump equipped with sufentanil injection will be connected,if the patient's resting NRS ≥ 4 points , they should be given sufentanil 5 ug intravenously at intervals of more than 8 minutes until NRS ≤ 3.
  Arms: LP group ：Nerve block with liposomal bupivacaine and intravenous analgesia group
Other: Intravenous analgesia — When the MOAA/S score is 5 after the surgery,the PCIA pump equipped with sufentanil injection will be connected,if the patient's resting NRS ≥ 4 points , they should be given sufentanil 5 ug intravenously at intervals of more than 8 minutes until NRS ≤ 3.
  Arms: control group：Intravenous analgesia group

SUMMARY:
To study the effectiveness of ACB and iPACK block with liposomal bupivacaine for postoperative analgesia in patients undergoing knee arthroplasty

DETAILED DESCRIPTION:
The pain after knee arthroplasty limits the patient's activities and postoperative recovery, and currently there are mainly three analgesic methods: intravenous analgesia, epidural analgesia and nerve block analgesia. There is a lack of studies on whether liposomal bupivacaine, if used for ACB and iPACK block, can achieve benefits in knee arthroplasty pain management by prolonging sensory nerve block without affecting muscle strength, improving patient prognosis, and shortening hospitalization days.

In this study, in order to better evaluate the effect of liposomal bupivacaine for ACB and iPACK biock on the prognosis of patients undergoing knee arthroplasty, not only the NRS and AUC of patients in each group will be observed, but also the postoperative QoR-15 Quality of Recovery Rating Scale, postoperative nausea, vomiting and other complications, and the number of hospitalization days will be also included as observation indicators. The completion of this study can provide a clinical basis for the selection of analgesic regimens for knee arthroplasty, and also provide strong evidence-based medical support for the relevant medical decision making of government departments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-79 years.
2. Patients undergoing unilateral total knee arthroplasty or unicondylar joint replacement.
3. Normal diet.
4. ASA grade I~Ⅲ;
5. BMI 18-30kg /m2.
6. No intraspinal anesthesia contraindications.

Exclusion Criteria:

1. Patients with severe neurological diseases.
2. Hearing and speech impaired.
3. Preoperative gastric emptying disorders, such as gastrointestinal obstruction, gastroesophageal reflux, or previous gastrointestinal surgery, etc.
4. Patients with severe renal insufficiency or other severe metabolic diseases.
5. Mental disorders, alcoholism or a history of drug abuse.
6. The surgical time is greater than 3 hours.
7. Puncture site infection, abnormal coagulation function, and local anesthetic allergy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The cumulative use of analgesic drugs (sufentanil,calculated in ug)up to 48 hours postoperative in each group | Up to 48 hours postoperative
  To study the effectiveness of ACB and iPACK block with liposomal bupivacaine for postoperative analgesia in patients undergoing knee arthroplasty.A lower dose of analgesics indicates a longer duration of block.

SECONDARY OUTCOMES:
NRS scores at rest and during exerciseat at 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours postoperative | at 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours postoperative
  The NRS typically consists of a straight line with numbers ranging from 0 to 10. Each number corresponds to a level of pain intensity:0: No pain.1 to 3: Mild pain （low intensity）. 4 to 6: Moderate pain （moderate intensity）. 7 to 10: Severe pain (high intensity) Patients are asked to choose a number that best represents their current pain level, where 0 means no pain, and 10 indicates the worst possible pain.A lower NRS score indicates a longer duration of block.
The total number of PCIA compressions on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Fewer total PCIA compressions indicated a longer duration of block.
The number of effective PCIA compressions on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Fewer total effective PCIA compressions indicated a longer duration of block.
The number of times of remedial analgesia on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Fewer times of rescue analgesia indicated a longer duration of analgesia.
The cumulative use of analgesic drugs (sufentanil,calculated in ug)on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Less cumulative use of analgesics indicates a longer duration of block
The percentage of subjects who did not use remedial analgesics on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  A greater percentage of subjects who did not use rescue analgesics indicated a longer duration of analgesic block.
Satisfaction score of subjects on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Rated on a 0-10 scale, with a higher score representing greater satisfaction.
Satisfaction score of surgeons on the first day,the second day and the third day after surgery. | On the first day,the second day and the third day after surgery.
  Rated on a 0-10 scale, with a higher score representing greater satisfaction.
Both the liposomal bupivacaine group and the ropivacaine group were subjected to ACB and iPACK block. Area under the pain intensity-time curve within 72 hours after the first postoperative dose(PI-AUC72)was observed in the three groups. | within 72 hours after the first postoperative initiation of drug administration
  A smaller PI-AUC72 indicates a longer duration of nerve block.
15-item Quality of Recovery Rating Scale (QoR-15): 24hours, 48hours and 72hours postoperatively | at 24 hours, 48 hours and 72 hours postoperative
  QoR-15 was used to assess five aspects of postoperative recovery quality (physical comfort, physical independence, psychological support, emotion and pain), with higher scores indicating the higher postoperative recovery quality. The lowest score is 0 points, and the highest score is 150 points.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Han, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kukreja P, Feinstein J, Kalagara HK, Huntley SR, Lee SR, Naranje S, Shah A. A Summary of the Anatomy and Current Regional Anesthesia Practices for Postoperative Pain Management in Total Knee Arthroplasty. Cureus. 2018 Jun 7;10(6):e2755. doi: 10.7759/cureus.2755. PMID 30094112
- [Background] Sundarathiti P, Ruananukul N, Channum T, Kitkunasathean C, Mantay A, Thammasakulsiri J, Sodsee W. A comparison of continuous femoral nerve block (CFNB) and continuous epidural infusion (CEI) in postoperative analgesia and knee rehabilitation after total knee arthroplasty (TKA). J Med Assoc Thai. 2009 Mar;92(3):328-34. PMID 19301724
- [Background] Fedriani de Matos JJ, Atienza Carrasco FJ, Diaz Crespo J, Moreno Martin A, Tatsidis Tatsidis P, Torres Morera LM. Effectiveness and safety of continuous ultrasound-guided femoral nerve block versus epidural analgesia after total knee arthroplasty. Rev Esp Anestesiol Reanim. 2017 Feb;64(2):79-85. doi: 10.1016/j.redar.2016.05.008. Epub 2016 Jul 9. English, Spanish. PMID 27400891
- [Background] Yu YL, Cao DH, Chen B, Yang ZH, You KZ. Continuous femoral nerve block and patient-controlled intravenous postoperative analgesia on Th1/Th2 in patients undergoing total knee arthroplasty. J Biol Regul Homeost Agents. 2018 May-Jun;32(3):641-647. PMID 29921393
- [Background] Vora MU, Nicholas TA, Kassel CA, Grant SA. Adductor canal block for knee surgical procedures: review article. J Clin Anesth. 2016 Dec;35:295-303. doi: 10.1016/j.jclinane.2016.08.021. Epub 2016 Oct 11. PMID 27871547
- [Background] Mou P, Wang D, Tang XM, Zeng WN, Zeng Y, Yang J, Zhou ZK. Adductor Canal Block Combined With IPACK Block for Postoperative Analgesia and Function Recovery Following Total Knee Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Study. J Arthroplasty. 2022 Feb;37(2):259-266. doi: 10.1016/j.arth.2021.10.004. Epub 2021 Oct 13. PMID 34653576
- [Background] Hasabo EA, Assar A, Mahmoud MM, Abdalrahman HA, Ibrahim EA, Hasanin MA, Emam AK, AbdelQadir YH, AbdelAzim AA, Ali AS. Adductor canal block versus femoral nerve block for pain control after total knee arthroplasty: A systematic review and Meta-analysis. Medicine (Baltimore). 2022 Aug 26;101(34):e30110. doi: 10.1097/MD.0000000000030110. PMID 36042669
- [Background] Hussain N, Brull R, Sheehy B, Dasu M, Weaver T, Abdallah FW. Does the addition of iPACK to adductor canal block in the presence or absence of periarticular local anesthetic infiltration improve analgesic and functional outcomes following total knee arthroplasty? A systematic review and meta-analysis. Reg Anesth Pain Med. 2021 Aug;46(8):713-721. doi: 10.1136/rapm-2021-102705. Epub 2021 May 14. PMID 33990436